CLINICAL TRIAL: NCT00616603
Title: The Effects of Dexamethasone on the Duration of Sciatic Nerve Blocks
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI is no longer here.
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 57164
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Results first posted 2014-06-11 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-06

CONDITIONS: Total Knee Arthroplasty
Keywords: Total Knee Arthroplasty.; Sciatic nerve Blocks.; Dexamethasone.
MeSH Terms: interventions — Ropivacaine; Dexamethasone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Other): This is the control arm and subjects in Group A will have sciatic nerve block with 20ml of 0.2% Ropivacaine + 2ml IV of normal saline.
  Interventions: Drug: Ropivacaine; Drug: Normal Saline
- Group B (Experimental): Subjects in Group B will have sciatic nerve block with 20ml of 0.2% Ropivacaine + 8mg Dexamethasone + 2ml IV of normal saline.
  Interventions: Drug: Ropivacaine; Drug: Dexamethasone; Drug: Normal Saline
- Group C (Active Comparator): Subjects in Group C will have sciatic nerve block with 20ml of 0.2% Ropivacaine + 2ml IV (8mg)of Dexamethasone.
  Interventions: Drug: Ropivacaine; Drug: Dexamethasone

INTERVENTIONS:
Drug: Ropivacaine — 20 ml of 0.2% ropivacaine injected locally as regional anesthesia given once.
Drug: Dexamethasone — 8mg Dexamethasone injected locally along with ropivacaine for regional anesthesia given once.
  Arms: Group B
Drug: Dexamethasone — 2ml(8mg)Dexamethasone given once intravenously.
  Arms: Group C
Drug: Normal Saline — 2ml of normal saline given once intravenously.
  Arms: Group A; Group B

SUMMARY:
Dexamethasone is a commonly used steroid. This medication has been used for many years by physicians for many different indications. Recent articles, multiple case reports, and experience at this institution have indicated that dexamethasone successfully prolongs the effective duration of local anesthetics for regional blocks. This can cause a significant reduction in postoperative pain and the decreased need for postoperative narcotics. Although other adjuncts can be used for prolonging nerve blocks, epinephrine causes local vasoconstriction which can cause ischemia and nerve damage in a large nerve such as the sciatic nerve.Dexamethasone will not cause this problem and yet could prolong the duration of a sciatic nerve block. Therefore, the goal of this study is to prospectively evaluate the effectiveness of dexamethasone, both locally through the nerve block and systemically via IV administration, in prolonging the effective duration of local anesthetics when used in sciatic nerve blocks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 yrs, male or female subjects.
* Subjects must be scheduled to undergo total knee arthroplasty under general anesthesia with consent for a femoral and sciatic nerve block post operatively for pain control.
* American Society of Anesthesiology Class 1,2,3,or 4.
* Capable of speaking and understanding English sufficiently to provide written informed consent and able to respond when asked.
* Weight > or equal to 60kg.

Exclusion Criteria:

* Any allergies or hypersensitivity to ropivacaine or dexamethasone.
* Subject is on chronic steroids preoperatively for any reason.
* History of chronic pain syndrome (i.e. CPRS, Lumbar radiculopathy).
* History of documented or stated nerve damage or neuropathy to the surgical lower extremity.
* Contraindication to placement of sciatic nerve block.
* Sciatic block placement failure.
* Subject mistakenly receives steroids intraoperatively.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2007-08; Primary Completion 2011-01 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Lee, MD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University Medical Center, Loma Linda, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment process began on 10/4/2007. The last subject to be recruited was on 02/23/2009. Subjects were consented at their Pre-anesthesia appointment or in the Observation Unit prior to their surgery.Some subjects were pre-consented by a resident on the phone prior to their surgery date.
Pre-assignment Details: We had 4 subjects withdraw because of screen failure, rescheduled surgery and physcian withdrawal.
Period: Overall Study
Arm/Group | Group A | Group B | Group C
Started | 14 | 14 | 15
Completed | 12 | 14 | 13
Not Completed | 2 | 0 | 2
Not completed — Physician Decision | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Total
Number analyzed (Participants) | 14 | 14 | 15 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 5 | 6 | 18
  >=65 years | 7 | 9 | 9 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.154 (10.597) | 67.692 (7.357) | 67.714 (7.859) | 65.525 (9.140)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 7 | 22
  Male | 6 | 7 | 8 | 21
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 15 | 43

OUTCOME MEASURES:

1. Primary Outcome: Duration of Sciatic Nerve Block
Description: Intraoperative opioid requirement PACU opioid requirement Floor opioid usage Time of onset of motor block (or weakness) Time of onset of sensory block Return of motor function Return of sensation Pain scores
Time Frame: from the time the block was placed up to 24 hours
Population: PI left the institution and no analysis completed due to questionable data integrity
Groups:
- Group A: This is the control arm and subjects in Group A will have sciatic nerve block with 20ml of 0.2% Ropivacaine + 2ml IV of normal sali
- Group B: Subjects in Group B will have 20ml of 0.2% Ropivacaine + 8mg Dexamethasone + 2ml of normal saline
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Description: Pi left institution and AEs were not assessed due to data integrity.
Arm/Group | Group B | Group A | Group C
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
PI left the institution and data analysis cannot be summarized due to poor data integrity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes